CLINICAL TRIAL: NCT01677884
Title: Intra-arterial Hepatic Bevacizumab and Systemic Chemotherapy in Hepatic Metastases of Metastatic Colorectal Cancer: a Phase II Multicentric Study With Patients in Progression After First Line Systemic Chemotherapy
Brief Title: Intra-arterial Hepatic Bevacizumab and Systemic Chemotherapy
Acronym: BEVIAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005559-15; CSET 2011/1827 (Other: Institut Gustave Roussy)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with metastatic CRC (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Irinotecan

INTERVENTIONS:
Drug: Bevacizumab — Every 3 weeks : 7.5 mg/kg intra arterial in 2 hours at D1
Drug: Capecitabine — Every 3 weeks: 2000 mg/m²/d in 2 times/d from D1 to D4
Drug: Irinotecan — Every 3 weeks: 200mg/m² in 30mn IV at D1 (if oxaliplatin in first line) or oxaliplatin 130mg/m² in 2h IV at D1 (if irinotecan in first line)

SUMMARY:
The purpose of the study is to assessed the efficiency of treatment based on the objective response rate (RECIST 1.1)

ELIGIBILITY:
Inclusion Criteria:

* Liver metastases of colon cancer or rectal predominant (histological evidence obtained on the primary tumor or liver metastases)

  * Isolated (no extra-hepatic metastasis, primary tumor resected)
  * No access to curative hepatectomy (R0 resection foreseeable or not leaving less than 30% residual non-tumor liver normally vascularized), or requiring complex hepatectomy, very large (5 or more segments) and / or risked (class II CPP)
  * which at least one measurable by RECIST (>2 cm, or >1 cm if Computed tomography (CT) spiraled)
  * Or extra-hepatic disease of small size potentially accessible to a resection (one or two lung metastases, lymphadenopathy localized accessible to curative resection)
  * colon or rectal primary tumor : resected or asymptomatic
* Progression after first line chemotherapy to treat the metastatic disease, all types of treatment allowed except intra-arterial Bevacizumab
* Age >18 years <75 years
* Performance status WHO 0 or 1
* Life expectancy >3 months
* Bilirubin <1.5 times the upper limit of normal (N), ASAT and ALAT <5N, creatinine <1.5 N neutrophils >1.5 x 10^9/L, platelets ≥100 x 10^9/L, hemoglobin >9g/dL. Patients may be included even if they were transfused
* CT (or MRI) reference for the measurement of metastases performed within 28 days before the first treatment cycle
* Information of the patient or legal representative signing the informed consent
* Affiliated to a social security system

Exclusion Criteria:

* Symptomatic colon or rectal primary tumor (sub-occlusion, significant hemorrhage, major rectal syndrome)
* Extra-hepatic metastases other than small size disease potentially accessible after resection
* Grade 3-4 allergy to one of the treatment compounds
* Two lines of prior chemotherapy. One line is allowed for metastatic disease but must have been started more than 6 months after completion of adjuvant treatment.
* Participation during or within 30 days before study to another therapeutic trial with an experimental molecule
* Concomitant cancer systemic treatment using immunotherapy, chemotherapy or hormone
* Symptomatic CHD or myocardial infarction within 6 months prior entry into the study, cardiac arrhythmia uncontrolled despite treatment
* Uncontrolled hypertension (blood pressure >150/100 mm Hg despite hypertensive treatment)
* Heart Failure >Grade II of the New York Heart Association (NYHA) (class II-III-IV)severe renal failure
* History and / or presence of bleeding disorders and/or thrombotic <6 months
* Uncontrolled Serious illness, uncontrolled active infection or other serious underlying condition which may prevent the patient to receive treatment
* Pregnancy (or positive pregnancy test at baseline), lactation or no contraception effective for men or women of childbearing age
* Occlusion or sub-bowel obstruction or history of inflammatory bowel disease
* Other cancer within 5 years prior to entry into the trial or concomitant (except in situ cancer of the cervix or skin basal-cell carcinoma properly treated)
* Legal inability (persons deprived of liberty or under guardianship)
* Inability to sign the consent or submit to medical test for geographical, social or psychological reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Efficiency of treatment based on objective response rate | Every 9 weeks from the start to tumoral progression

SECONDARY OUTCOMES:
Treatment toxicity based on NCI-CTC v4.0 | Every 3 weeks from the start to tumoral progression or toxicity preventing further processing
Progression Free Survival | Every 9 weeks form the start to tumoral progression
Hepatic metastasis resection rate | Assessed up 6 months after the end of treatment

OTHER OUTCOMES:
Total area under the curve of contrast-enhanced liver ultrasound | Assessed up in baseline, D7, D14, W4, W7 and every 9 weeks up to progression

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ducreux, MD-PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, Val de Marne, France